CLINICAL TRIAL: NCT03297957
Title: Evaluation of Fluorescence Imaging in Head and Neck Cancer
Brief Title: Fluorescence Imaging in Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201708068
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Cancer; Cancer of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1: Goggle Imaging (Experimental): -Patient will then be taken to the operating room for this surgical procedure. Prior to starting the operation, the patient will undergo injection of ICG around the tumor per standard techniques while in the operating room. Those undergoing intraoperative visualization of parathyroid glands will not have any administration of ICG as these glands autofluoresce. Patients will then undergo the standard SLN biopsy procedure (those undergoing parathyroid visualization will not undergo this). The surgeon will put on the goggle system to attempt to identify the SLN using fluorescence guidance or parathryroid visualization. After this is performed, the goggle system will be removed and the procedure will be completed per normal.
  Interventions: Device: Hands-free goggle system

INTERVENTIONS:
Device: Hands-free goggle system — -Manufactured at Washington University

SUMMARY:
Fluorescent technology continues to advance in the detection of sentinel lymph nodes (SLNs). Currently, this requires switching from near-infrared light to white light to be able to identify the fluorescent tissue contrasting with normal surrounding tissue. Currently, no system has been studied specifically for head and neck sentinel lymph node biopsies using a hands free goggle system that can visualize white light (normal surgical visualization) and nearinfrared light (ICG fluorescence) simultaneously. This technology may have implications on the safety and accuracy of sentinel lymph node biopsy for head and neck mucosal and cutaneous tumors. Secondarily, this may reduce operative costs by decreasing the amount of time required to perform the SLNB procedure.

Regarding parathyroid identification, this technology has the potential to identify these very small glands during procedures they are at risk. These glands are not only at risk of inadvertent removal if not adequately identified, but may also be at risk if devascularized by manipulation during the surgical procedure. Therefore, early and accurate identification may decrease the rate of temporary and permanent hypoparathyroidism and hypocalcemia. This is not only an issue during thyroid and parathyroid surgery, but during laryngectomy surgery where the anatomic region these glands are located are often resected to remove at risk lymph nodes from cancer spread. Therefore, identifying these glands may help preserve parathyroid function in this patient population as well.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older will be considered eligible.
* Patients with head and neck malignancies, such as melanoma, non-melanoma cutaneous malignancies, or oral cavity squamous cell carcinoma. Patients with central neck pathology including thyroid neoplasms, parathyroid neoplasms, and laryngeal neoplasms undergoing surgical resection.

  * Candidates for sentinel lymph node biopsy or central neck surgery
  * Newly diagnosed with clinically node negative head and neck cancer being staged with sentinel lymph node biopsy.
* Not pregnant or breast feeding.
* Able to understand and willing to sign an IRB-approved written informed consent document.
* Able to understand written or spoken English.

Exclusion Criteria:

* History of allergy to iodide drugs or shellfish (iodine allergy)
* Pregnant or breast feeding
* Do not fit age criteria
* Prisoners
* Unable to provide written consent
* Contraindications for surgery

  *Presence of uncontrolled intercurrent illness including, but not limited to, ongoing or active infection of the head and neck, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of using a novel fluorescence imaging device to detect a SLN as measured by the ability of the imaging device to identity the SLN by the surgeon during the standard biopsy procedure | Up to 1 week after surgery
  -Feasibility will be assessed in terms of percentage of patients enrolled for whom peri-tumoral injection with ICG is performed successfully
Feasibility of using a novel fluorescence imaging device to detect a SLN as measured by the ability of the imaging device to identity the SLN by the surgeon during the standard biopsy procedure | Up to 1 week after surgery
  -Feasibility will be assessed in terms of percentage patients whom the sentinel and superficial lymph nodes will be detected from the hands free goggle device
Feasibility of using a novel fluorescence imaging device to detect a SLN as measured by the ability of the imaging device to identity the SLN by the surgeon during the standard biopsy procedure | Up to 1 week after surgery
  -Feasibility will be assessed in terms of percentage of total lesions identified from the new technique are truly positive as confirmed by biopsy
Feasibility of using a novel fluorescence imaging device to detect a SLN as measured by the ability of the imaging device to identity the SLN by the surgeon during the standard biopsy procedure | Up to 1 week after surgery
  -Feasibility will be assessed in terms of the the percentage of total positive SNLs being missed from the new device
Ability of the hands-free goggle system to identify parathryoid glands during central neck surgeries | Up to 1 week after surgery

SECONDARY OUTCOMES:
Determine if there is contrast between SLN and surrounding tissues using the novel fluorescence imaging device | Up to 1 week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ryan S Jackson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu